CLINICAL TRIAL: NCT04848493
Title: A National, Multicentric, Observational, Prospective Study to Assess Immune Response to COVID-19 Vaccine in Frail Patients (VAX4FRAIL).
Brief Title: National Project on Vaccines, COVID-19 and Frail Patients
Acronym: VAX4FRAIL
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Istituto Clinico Humanitas (Other); IRCCS San Raffaele (Other); Regina Elena Cancer Institute (Other); Istituto Nazionale per le Malattie Infettive "Lazzaro Spallanzani" IRCCS (Network); University of Roma La Sapienza (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Istituti Fisioterapici Ospitalieri (Other); Istituto Tumori Giovanni Paolo II, BARI (Unknown); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: VAX4FRAIL study
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: COVID-19; Solid Tumor; Hematologic Diseases; Neurologic Disorder; Rheumatic Diseases
Keywords: vaccination; COVID-19; frail patients
MeSH Terms: conditions — COVID-19; Hematologic Diseases; Nervous System Diseases; Rheumatic Diseases | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anti-spike SARS-CoV-2 S1/S2 IgG (CE mark, part number 311450)
  * Anti-N SARS-CoV-2 IgG (CE mark, 6R86-22).
  * Neutralization Whole blood cell-mediated immunity assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- HEMATOLOGICAL MALIGNANCIES: 1a. Newly diagnosed patients with ANY haematological malignancy requiring treatment (No.=100).
  1b. Patients with ongoing treatments or with treatments completed within 6 months (chemotherapy and target therapies) other than antibodies. More specifically: patients with ongoing or completed chemotherapy (No.=50) or patients with ongoing or completed Ibrutinib (No.=50) or patients with ongoing or completed ruxolitinib (No.=50)
  1c. Patients treated with anti-CD19 or CD20 or CD22 or CD30 or anti-PD1 antibodies with or without chemotherapy OR patients receiving CAR-T cells: patients treated anti-B-cell (No.=50) or patients treated anti-CD30 (No.=50) or patients treated anti-PD1 (No.=50).
  1d. Patients at three months after autologous or allogeneic transplantation without active immune suppressive therapy: after autologous transplantation (No.=50) or after allogenic transplantation (No.=50).
  Interventions: Biological: COVID-19 vaccines
- SOLID TUMORS: 2a. Chemotherapy in adjuvant therapy. All patients with a diagnosis of solid tumors apart resected basal-cell or squamous-cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, and carcinoma in situ of the Breast. Under curative surgery (stage II-III) for the solid tumor or hemotherapy alone or in combination with target therapies or radiotherapy (No.=100).
  2b. Chemotherapy in metastatic Disease. All patients with a diagnosis of solid tumors with Metastatic disease (stage IV), undergoing chemotherapy alone or in combination with immunotherapy or target therapy (No.=100).
  2c. Immunotherapy in metastatic Disease. All patients with a diagnosis of solid tumors with Metastatic disease (stage IV), undergoing immunotherapy alone (No.=100).
  2d. Target therapies in metastatic Disease. All patients with a diagnosis of solid tumors with Metastatic disease (stage IV), Undergoing target therapy alone (No.=100)
  Interventions: Biological: COVID-19 vaccines
- IMMUNORHEUMATOLOGICAL DISEASES: 3a. Patients with ANCA-associated vasculitis classified according to Chapel Hill Consensus Conference nomenclature, treated with immunodepressants agents with/without glucocorticoids (No.=50) or treated with RTX with/without glucocorticoids (No.=50) 3b. Interstitial Lung Disease in Autoimmune Conditions. Patients with a diagnosis of a specific CTD, myositis or rheumatoid arthritis based on validated classification criteria, and clinically significant ILD defined as disease treated with traditional immunodepressants or rituximab and fibrotic and/or inflammatory changes on chest CT not attributable to infection, and no evidence of obstructive lung disease. Patients treated with traditional immunodepressive agents with/without glucocorticoidspatients (No.=50) or patients treated with rituximab with/without glucocorticoids (No.=50)
  Interventions: Biological: COVID-19 vaccines
- NEUROLOGICAL DISEASES: 4a. Patients with a diagnosis of multiple sclerosis, age < 60 years with relapsing-remitting MS on Ocrelizumab (anti-CD20 monoclonal antibody) (No.=50) or with secondary/primary progressive MS on Ocrelizumab (anti-CD20 monoclonal antibody) (No.=50).
  4b. Generalized Myasthenia Gravis, on immunosuppressive polytherapies or on B-cell targeted biological treatments, with lymphocytes count < 1 cell/microliter, or with thymoma (No.=100)
  Interventions: Biological: COVID-19 vaccines

INTERVENTIONS:
Biological: COVID-19 vaccines — This is an observational prospective study whose general objective is to assess the impact of COVID-19 vaccination in terms of induction of humoral and cell-mediated immune responses in selected fragile (altered immunocompetence) populations.

SUMMARY:
This is a multicentre observational study with the aim of evaluating the antibody and cellular response after vaccination for SARS-CoV-2 with Pfizer-BioNTech or Moderna vaccines in frail subjects with impaired immuno-competence, due to their underlying diseases or ongoing therapies.

DETAILED DESCRIPTION:
The immune response to COVID-19 vaccination will be assessed at the following time points:

T0: the day of vaccination T1: the day of the booster dose according to the schedule of the two vaccines (Pfizer/BioNTech or Moderna) T2: between 5 and 7 weeks after T0 for those vaccinated with Pfizer/BioNTech and between 6 and 8 weeks after T0 for those vaccinated with Moderna.

* T3: 12 (± 1) weeks after T0
* T4: 24 (± 2) weeks from T0
* T5: 52 (± 2) weeks from T0 Prevention of SARS-CoV-2 infection will be assessed in terms of incidence of SARS-CoV-2 infections (NF molecular swab positive), and of SARS-CoV-2 infections requiring hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Any subject undergoing SARS-CoV-2 vaccination with Pfizer-BioNTech or Moderna vaccines may be included in the study if they belong to at least one of the subgroups listed below:

  1. Hematological tumors
  2. Solid tumors
  3. Rheumatological diseases
  4. Neurological diseases

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any subject undergoing SARS-CoV-2 vaccination can be enrolled in the study if included in at least one of the below subgroups due to the proper underlying conditions:
  HEMATOLOGICAL MALIGNANCIES These subgroups have been decided considering that patients with hematological malignancies have a low immune response because of the lympholytic treatment they receive.
  SOLID TUMORS (2). ANCA-associated vasculitis Interstitial lung disease (ILD) is a feature of many connective tissue diseases (CTDs), including systemic sclerosis, mixed connective tissue disease, systemic lupus erythematosus, and Sjogren syndrome, of dermatomyositis and polymyositis, and of rheumatoid arthritis.
  Multiple sclerosis
  Generalized Myasthenia Gravis Patients with myasthenia gravis
Sampling Method: Non-Probability Sample
Enrollment: 747 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 vaccine immunization | 5-7 weeks after T0 for Pfizer/BioNTech vaccination; 6-8 weeks after T0 for Moderna vaccination
  For assessing the immunologic response to the COVID-19 vaccination, the anti-S antibodies levels in the fragile population will be quantified at T2 and compared with the anti-S antibodies levels quantified at the same time point in a population of healthy subjects.

SECONDARY OUTCOMES:
anti-S antibodies immunological response | at 6 times points T0 before vaccine administration, T1 before the second dose of the vaccine and at times T2, T3, T4 and T5 which correspond to 5-7 weeks (Pfizer-BioNTech) or 6-8 weeks (Moderna), 12 weeks, 24 weeks and 52 weeks after the first dose
  for each time point, the anti-S antibodies levels will be quantified and compared with the anti-S antibodies levels quantified at the same time point in a population of healthy subjects (see controls).
T cell immunological response | at 6 times points T0 before vaccine administration, T1 before the second dose of the vaccine and at times T2, T3, T4 and T5 which correspond to 5-7 weeks (Pfizer-BioNTech) or 6-8 weeks (Moderna), 12 weeks, 24 weeks and 52 weeks after the first dose
  At each time point, the Spike and N-specific T-cell immunity of the 1300 enrolled subjects will be assessed and compared to that observed in a population of healthy subjects at the same time point (see controls).
immunological response in different subgroups | 1 year
  Subgroup analysis on the immunological response will be performed according to the clinical characteristics of the patients, the main diagnosis subgroups according to the eligibility criteria and the treatments they have received. we will compare the immune response with the different clinical characteristics of the patients
impact of COVID-19 vaccination on patient health status | 1 weeks after frist dose and 1 week after second dose
  The impact on health status will be assessed through a questionnaire compiled at T1 and T2 by the physician before the blood sampling. The questionnaire will assess the occurrence of a list of symptoms in the week after the first and second administration of the vaccine.
incidence of SARS-CoV-2 infection. | all 52 weeks
  The incidence of SARS-CoV-2 infection will be assessed in terms of number and proportion of patients who during the 52 weeks. SARS-CoV-2 infection will be assessed with: positive to molecular NF swab.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Salvarani, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (12):
- Italy (12):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari, Bari
  - IRCCS Azienda Ospedaliera Universitaria, Bologna, Bologhna
  - Ospedale Policlinico San Martino IRCCS, Genova, Genova
  - Foindazione IRCCS Istituto Neurologico Carlo Besta, Milan, Milano
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milano
  - IRCCS Istituto Clinico Humanitas, Milan, Milano
  - IRCCS Ospedale San Raffaele, Milan, Milano
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Reggio Emilia
  - IRCCS Istituto Nazionale Tumori Regina Elena, Roma, Roma
  - IRCCS Istituto per le Malattie Infettive Lazzaro Spallanzani, Roma, Roma
  - Istituto Dermatologico San Gallicano, Roma, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Cosimo S, Lupo-Stanghellini MT, Costantini M, Mantegazza R, Ciceri F, Salvarani C, Zinzani PL, Mantovani A, Ciliberto G, Uccelli A, Baldanti F, Apolone G, Delcuratolo S, Morrone A, Locatelli F, Agrati C, Silvestris N. Safety of third dose of COVID-19 vaccination in frail patients: Results from the prospective Italian VAX4FRAIL study. Front Oncol. 2022 Oct 20;12:1002168. doi: 10.3389/fonc.2022.1002168. eCollection 2022. PMID 36338743